CLINICAL TRIAL: NCT06811532
Title: Assessing Perfusion of an Osteotomised Scapula and Latissimus Dorsi Chimeric Free Flap on the Thoracodorsal Artery
Brief Title: Assessing Perfusion of Osteotomized Scapula and Lat Flap
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Danielle MacNeil, Principal Investigator, Western University, Canada
Other Study IDs: 126223
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; scapular free flap; blood perfusion
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Blood perfusion analysis using SPY-Q software — Use of the SPY-Q analysis software during surgery to calculate bone profusion scores on several areas of the scapular tip flap (endosteum of scapula bone segments and latissimus dorsi muscle component).

SUMMARY:
The gold standard for reconstruction of the jaw is the utilization of a bone free tissue transfer. Scapula reconstruction is an excellent option for elderly patients, those with significant comorbidities and for complex defects with large soft tissue reconstructive requirements. The scapula is supplied by the angular artery and circumflex scapula arteries. No studies have shown with objective measures, the viability of the lateral border of the scapula bone supplied by either the angular artery or circumflex scapula arteries. The aim of this observational study is to demonstrate with objective clinical measures, via SPY-Q software analysis, that the angular artery can adequately supply the scapula tip flap including with a single osteotomy giving two bone segments, in 30 patients who will undergo reconstructive head and neck surgery at LHSC.

DETAILED DESCRIPTION:
The aim of this follow-up observational study is to demonstrate with objective clinical measures via SPY-Q software analysis, that the angular artery can adequately supply the scapula tip flap including a single distal osteotomy segment. 30 patients undergoing mandible or maxillary reconstruction with the scapular tip flap will be included. An osteotomy will be performed at up to 8cm from the scapular tip. The adequacy of blood supply to the scapula tip flap after a distal osteotomy and the latissimus dorsi muscle component of the flap will be measured intraoperatively, using SPY-Q software analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (18 years and older) seen at the head and neck clinic at London Health Sciences Centre (LHSC)

  * Planned to undergo a maxillary and/or mandibular reconstruction surgery with a scapular tip flap

Exclusion Criteria:

* • Younger than 18 years of age

  * History of failing microvascular flaps
  * Hypersensitivity toward ICG or related substances (e.g., imaging agents), defined as (based on ICG product monograph): possibly life-threatening dizziness, severe itching, hives, nausea, difficulty breathing, rash, low blood pressure)
  * Pregnant
  * Breastfeeding
  * Clinically apparent cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced head and neck cancer, benign tumors of the jaw and osteoradionecrosis, scheduled for head and neck reconstructive surgery using the scapular tip flap at London Health Sciences Centre (LHSC).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-07 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Adequacy of blood perfusion of osteomized lateral border of the scapula bone supplied by the angular artery | Intra-operatively
  To measure the adequacy of blood perfusion of osteotomised lateral border of the scapula bone supplied by the angular artery via SPY-Q analysis in patients undergoing a scapular tip flap for reconstruction of a jaw defect
Blood perfusion of osteomized lateral border of the scapula | Intra-operatively
  To measure the adequacy of blood perfusion of osteotomised lateral border of the scapula bone supplied by the angular artery via SPY-Q analysis in patients undergoing a scapular tip flap for reconstruction of a jaw defect

SECONDARY OUTCOMES:
To assess flap viability | Intra-operatively; up to 10 days post-operatively
  To evaluate whether scapular tip flaps with an osteotomy with adequate bone perfusion scores resulted in surgical success (flap viability)
Concordance between subjective and objective measure of blood perfusion | Intra-operatively; up to 10 days post-operatively
  To assess the concordance between visual inspection of blood perfusion and SPY-Q analysis of blood perfusion
Blood perfusion of latissmus dorsi | Intra-operatively
  To measure the adequacy of blood perfusion of the latissimus dorsi muscle component of the scapula flap via SPY-Q analysis

CONTACTS AND LOCATIONS:
Overall Officials: Danielle MacNeil, MD, Principal Investigator — Department of Otolaryngology-Head & Neck Surgery, Western University Canada

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request